CLINICAL TRIAL: NCT02805153
Title: The Multi-center, Open-label,Randomized Comparison Phase IV Clinical Trial of Efficacy and Safety of PEG-rhG-CSF in Preventing Neutropenia in Patients With Breast Cancer Receiving Chemotherapy
Brief Title: PEG-rhG-CSF in Patients With Breast Cancer Receiving Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSPC-PGC-IV-01
Record Dates: First submitted 2016-06-13; First posted 2016-06-17 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: PEG-rhG-CSF
MeSH Terms: conditions — Breast Neoplasms | interventions — pegylated granulocyte colony-stimulating factor; pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental/PEG-rhG-CSF (Experimental): patients received a single dose of 100 ug/kg of PEG-rhG-CSF(pegfilgrastim), on the basis of actual body weight, as a single subcutaneous injection on day 3 after chemotherapy.
  Interventions: Drug: PEG-rhG-CSF
- Active Comparator/rhG-CSF (Active Comparator): patients received daily subcutaneous injections of rhG-CSF(filgrastim) 5 ug/ kg/day. Injections on day 3 after chemotherapy and continued daily until an ANC of at least 10.0 X 10^9/L was documented after the expected nadir, or for a maximum of 14 days
  Interventions: Drug: rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF
  Other Names: pegfilgrastim
  Arms: Experimental/PEG-rhG-CSF
Drug: rhG-CSF
  Other Names: filgrastim
  Arms: Active Comparator/rhG-CSF

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PEG-rhG-CSF in patients with breast cancer receiving chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 and 70 years
* diagnosis of breast cancer patients
* chemotherapy naive
* Karnofsky Performance Status ≥ 70
* Written informed consent are acquired

Exclusion Criteria:

* uncontrolled infection
* Have accepted radiotherapy within 4 weeks before anticipated the study
* pregnancy
* Other situations that investigators consider as contra-indication for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
the occurrence rate of grade IV neutropenia during the first chemotherapy cycle | through first cycle of chemotherapy,an average of 1 month

SECONDARY OUTCOMES:
the non-occurrence rate of grade IV neutropenia (ANC < 0.5 x 10^9/L)during the next three consecutive cycles chemotherapy(except the first chemotherapy cycle) | through the next three consecutive cycles chemotherapy,an average of 3 months
the duration of grade IV neutropenia (ANC < 0.5 x 10^9/L) during the next three consecutive cycles chemotherapy(except the first chemotherapy cycle) | through the next three consecutive cycles chemotherapy,an average of 3 months